CLINICAL TRIAL: NCT05723601
Title: Addressing Preference as a Patient-centered Outcome to Prevent Recurrent Urinary Tract Infection (rUTI) in Post-menopausal Women: a Cross-over Randomized Controlled Trial
Brief Title: Preference of Women With Recurrent Urinary Tract Infection for Vaginal Estradiol Tablet vs Cream
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00092892
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Urinary Tract Infection
Keywords: vaginal estradiol cream; vaginal estradiol tablet
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- cream used first and then switch to tablets (Active Comparator): participants will start with 3 months of cream and then switch to tablets
  Interventions: Drug: Estradiol vaginal cream; Drug: Estradiol Vaginal Tablet
- tablets used first and switch to cream (Active Comparator): participants will start with 3 months of tablets and switch to cream
  Interventions: Drug: Estradiol vaginal cream; Drug: Estradiol Vaginal Tablet

INTERVENTIONS:
Drug: Estradiol vaginal cream — Participants will use vaginal estradiol cream for 3 months
Drug: Estradiol Vaginal Tablet — Participants will use vaginal estradiol tablet for 3 months

SUMMARY:
Vaginally applied estrogen has been shown to decrease the incidence of Recurrent Urinary Tract Infection (rUTI) in post-menopausal women. However, prior studies have shown the compliance rate for topical estrogen cream is low. The vaginal estradiol tablet has been shown to be preferred by patients being treated for genitourinary syndrome of menopause and has improved compliance. There are no studies looking at the preference of post-menopausal women with rUTI for vaginal estradiol tablet as an alternative to vaginal estradiol cream.

DETAILED DESCRIPTION:
This study is a cross-over randomized study to assess preference. Participants will be in the study for 6 months, they will use vaginal estradiol cream for 3 months and vaginal estradiol tablet for 3 months. Patients who meet diagnostic criteria for rUTI will be recruited. Group A participants will start with 3 months of cream and then switch to tablets. Group B will start with 3 months of tablets and switch to cream. In addition, participants may be started on other supplemental medications (Cranberry, D-mannose, methenamine) at the discretion of their provider. Patients will get monthly phone calls to assess for side effects, safety concerns, and symptoms of UTI.

ELIGIBILITY:
Inclusion Criteria:

* Women age 20-80 who are post-menopausal or have undergone surgical menopause. Post-menopausal defined as amenorrhea for ≥ 1 year, or surgical menopause through bilateral oophorectomy, or menopausal symptoms for ≥ 1 year in women with prior hysterectomy
* New or previous diagnosis of recurrent Urinary Tract Infections (rUTI) (3 or more UTIs in the past year or 2 or more UTIs in the last 6 months) Must have at least one culture documented UTI, the remaining can be documented by urinalysis showing nitrites and leukocyte esterase.
* Not currently taking daily prophylactic antibiotics
* Willing to use vaginal estrogen for prevention of recurrent UTIs

Exclusion Criteria:

* Interstitial cystitis or bladder pain syndrome, nephrolithiasis, genitourinary abnormalities, fistula, history of renal transplant or anatomic abnormality of the kidney
* Fecal incontinence, intermittent catheterization or indwelling catheter, poorly controlled DM, urothelial cancer, estrogen-sensitive cancer including active breast cancer
* Recent urologic surgery within 3 months
* Inability to retain vaginal tablet (ex due to advanced prolapse, history of colpocleisis)
* Other medical reasons that are deemed incompatible with vaginal estrogen treatment
* Use of vaginal estrogen in the past 1 month- patients can be recruited after a 1 month wash-out period
* Inability to follow up at clinic study site to give sample, for example due to transportation issues
* Organ transplant patients
* Patients on systemic hormone replacement therapy (HRT)

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 21 (Actual)
Dates: Start 2024-01-12 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Patient preference rate for vaginal estradiol cream versus tablet | month 6
  Preference will be assess at 6 months or at the time of withdrawal, by asking participants: "Which route of vaginal estrogen do you prefer: Vaginal estradiol tablet or vaginal estradiol cream?"

SECONDARY OUTCOMES:
Change in vaginal and urinary microbiome Lactobacillus amount with the use of vaginal estradiol tablet versus cream | Baseline, Month 3, and Month 6
  Vaginal culture swab and urine culture specimens will be collected - The specimens will be sent for species-specific polymerase chain reaction (PCR) for Lactobacillus
Change in overall satisfaction, convenience, side effects, and effectiveness of vaginal estradiol cream vs tablet using Treatment Satisfaction Questionnaire for Medication (TSQM) | Month 3 and Month 6
  Treatment Satisfaction Questionnaire for Medication (TSQM) - The TSQM domain scores range from 0 to 100 with higher scores representing higher satisfaction on that domain. A questionnaire assessing adherence and the reasons for not taking drug at the recommended frequency of administration.
Changes in adherence scores | Month 3 and Month 6
  Adherence will be assessed by the medication adherence questionnaire (MAQ) - The MAQ will be used to determine medication adherence. This questionnaire asks respondents about past experience in taking medications. The responses are 'yes' or 'no' and are scored as yes=1 and no=0. Scores will be summed: high adherence = score of 0 points; medium adherence = score of 1-2 points, and low adherence = score of 3-4 points. Means and standard deviations will be compared within and between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Candace Parker-Autry, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No data will be shared with other researchers

REFERENCES:
- [Background] Walters, M.D. and M.M. Karram, Urogynecology and Pelvic Reconstructive surgery. 2022: Mosby Elsevier.
- [Background] Minkin MJ, Maamari R, Reiter S. Improved compliance and patient satisfaction with estradiol vaginal tablets in postmenopausal women previously treated with another local estrogen therapy. Int J Womens Health. 2013;5:133-9. doi: 10.2147/IJWH.S41897. Epub 2013 Mar 15. PMID 23526171
- [Background] Ferrante KL, Wasenda EJ, Jung CE, Adams-Piper ER, Lukacz ES. Vaginal Estrogen for the Prevention of Recurrent Urinary Tract Infection in Postmenopausal Women: A Randomized Clinical Trial. Female Pelvic Med Reconstr Surg. 2021 Feb 1;27(2):112-117. doi: 10.1097/SPV.0000000000000749. PMID 31232721
- [Background] Raz R, Stamm WE. A controlled trial of intravaginal estriol in postmenopausal women with recurrent urinary tract infections. N Engl J Med. 1993 Sep 9;329(11):753-6. doi: 10.1056/NEJM199309093291102. PMID 8350884
- [Background] Boris S, Suarez JE, Vazquez F, Barbes C. Adherence of human vaginal lactobacilli to vaginal epithelial cells and interaction with uropathogens. Infect Immun. 1998 May;66(5):1985-9. doi: 10.1128/IAI.66.5.1985-1989.1998. PMID 9573080
- [Background] O'Hanlon DE, Moench TR, Cone RA. Vaginal pH and microbicidal lactic acid when lactobacilli dominate the microbiota. PLoS One. 2013 Nov 6;8(11):e80074. doi: 10.1371/journal.pone.0080074. eCollection 2013. PMID 24223212
- [Background] Anger J, Lee U, Ackerman AL, Chou R, Chughtai B, Clemens JQ, Hickling D, Kapoor A, Kenton KS, Kaufman MR, Rondanina MA, Stapleton A, Stothers L, Chai TC. Recurrent Uncomplicated Urinary Tract Infections in Women: AUA/CUA/SUFU Guideline. J Urol. 2019 Aug;202(2):282-289. doi: 10.1097/JU.0000000000000296. Epub 2019 Jul 8. PMID 31042112
- [Background] Suckling J, Lethaby A, Kennedy R. Local oestrogen for vaginal atrophy in postmenopausal women. Cochrane Database Syst Rev. 2006 Oct 18;(4):CD001500. doi: 10.1002/14651858.CD001500.pub2. PMID 17054136
- [Background] Eriksen B. A randomized, open, parallel-group study on the preventive effect of an estradiol-releasing vaginal ring (Estring) on recurrent urinary tract infections in postmenopausal women. Am J Obstet Gynecol. 1999 May;180(5):1072-9. doi: 10.1016/s0002-9378(99)70597-1. PMID 10329858
- [Background] Weissmann-Brenner A, Bayevsky T, Yoles I. Compliance to vaginal treatment-tablets versus cream: a retrospective 9 years study. Menopause. 2017 Jan;24(1):73-76. doi: 10.1097/GME.0000000000000729. PMID 27648663
- [Background] Ventola CL. The antibiotic resistance crisis: part 1: causes and threats. P T. 2015 Apr;40(4):277-83. PMID 25859123
- [Background] Dason S, Dason JT, Kapoor A. Guidelines for the diagnosis and management of recurrent urinary tract infection in women. Can Urol Assoc J. 2011 Oct;5(5):316-22. doi: 10.5489/cuaj.11214. No abstract available. PMID 22031610
- [Background] Morisky DE, Green LW, Levine DM. Concurrent and predictive validity of a self-reported measure of medication adherence. Med Care. 1986 Jan;24(1):67-74. doi: 10.1097/00005650-198601000-00007. PMID 3945130
- [Background] Atkinson MJ, Sinha A, Hass SL, Colman SS, Kumar RN, Brod M, Rowland CR. Validation of a general measure of treatment satisfaction, the Treatment Satisfaction Questionnaire for Medication (TSQM), using a national panel study of chronic disease. Health Qual Life Outcomes. 2004 Feb 26;2:12. doi: 10.1186/1477-7525-2-12. PMID 14987333
- [Background] Rioux JE, Devlin MC, Gelfand MM, Steinberg WM, Hepburn DS. 17beta-estradiol vaginal tablet versus conjugated equine estrogen vaginal cream to relieve menopausal atrophic vaginitis. Menopause. 2018 Nov;25(11):1208-1213. doi: 10.1097/GME.0000000000001220. PMID 30358715